CLINICAL TRIAL: NCT00937794
Title: A Screening Study to Identify Pediatric Patients With Hunter Syndrome Who Demonstrate Evidence of Central Nervous System Involvement and Who Are Currently Receiving Treatment With Elaprase®
Brief Title: Screening Study to Identify Pediatric Patients With Hunter Syndrome Who Demonstrate Evidence of Central Nervous System (CNS) Involvement and Who Are Currently Receiving Treatment With Elaprase®
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: HGT-HIT-050
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Hunter Syndrome
MeSH Terms: conditions — Mucopolysaccharidosis II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: This is a screening study designed to evaluate the behavioral, physical, and neurodevelopmental status in pediatric patients with Hunter syndrome who have early signs and symptoms of CNS involvement and who are currently receiving treatment with Elaprase.
  Interventions: Behavioral: Neurobehavioral testing; Other: Visual and auditory assessments

INTERVENTIONS:
Behavioral: Neurobehavioral testing — If the patient is found to be eligible after completion of a telephone interview, he will undergo further testing to assess his neurodevelopmental status using a standardized battery of neurobehavioral testing.
Other: Visual and auditory assessments — If the patient is found to be eligible after completion of a telephone interview, he will undergo further testing to evaluate his visual and auditory function.

SUMMARY:
This study is being conducted to identify pediatric patients with Hunter syndrome who have neurodevelopmental disease characteristics, who are currently receiving treatment with Elaprase, and who may be suitable to participate in a clinical study with an investigational agent.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is male and is ≥3 and <18 years of age
2. The patient is currently receiving weekly IV infusions of Elaprase.
3. The patient, patient's parent(s), or legally authorized guardian(s) has voluntarily signed an Institutional Review Board / Independent Ethics Committee-approved informed consent form after all relevant aspects of the study have been explained and discussed with the patient. The guardians' consent and subject's assent, as relevant, must be obtained.

Exclusion Criteria:

1. The patient has a CNS shunt.
2. The patient has received a hematopoietic stem cell transplant.
3. The patient is currently enrolled in a clinical trial.
4. The patient has a significant medical or psychiatric comorbidity(ies) that might affect study data or confound the integrity of study results.

Ages: 32 Months to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Initial patient eligibility will be based on patient age and gender. Patients must be receiving weekly IV Elaprase infusions to be eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2009-07-02 (Actual); Primary Completion 2011-07-13 (Actual); Study Completion 2011-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States
- Birmingham Children's Hospital, Birmingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This screening study evaluated patients for disease and neurodevelopmental status to determine their potential eligibility for investigational study HGT-HIT-045 (NCT00920647), and informed decisions regarding study design, rate of enrollment, and estimated dates of completion for subsequent investigational studies in Hunter syndrome.
Groups:
- All Patients: All patients who met the inclusion criteria and consented to participate in the study.
Period: Overall Study
Arm/Group | All Patients
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.42 (2.841)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 33
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21
  United Kingdom | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Screened For The Follow-On Study With an Investigational Agent
Description: Standardized tests were used to identify patients who were receiving treatment with Elaprase, had cognitive impairment, and were suitable to participate in the follow-on clinical study (HGT-HIT-045). Assessments included: 1-Cognition: The Differential Ability Scale, Second Edition (DAS-II) or the Bayley Scales of Infant Development, Third Edition (BSID-III); 2-Adaptive Behavior: The Scale of Independent Behavior-Revised (SIB-R); 3-Executive Function: The Behavior Rating Inventory of Executive Function-Preschool version (BRIEF-P) for children or the Behavior Rating Inventory of Executive Function (BRIEF) for children less than or ≥6 years of age, respectively; 4-Motor: The Peabody Developmental Motor Scales-2 (PDMS-2) or the Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2) for children less than or ≥6 years of age, respectively.
Time Frame: 1 month
Population: All enrolled patients, defined as patients who met the inclusion criteria and consented to participate in the study.
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 33
participants | 17

2. Primary Outcome: Number of Participants With a Score of at Least 90 on The General Conceptual Ability (GCA) Sub-Scale of The Differential Ability Scale (DAS)
Description: The GCA sub-scale of the DAS, Second Edition (DAS-II) was used to obtain a general measure of cognitive ability.The maximum score is 120, with a higher score indicating greater cognitive ability. A score of 100 is considered an average score.
Time Frame: 1 month
Population: All enrolled patients, defined as patients who met the inclusion criteria and consented to participate in the study.
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 33
participants | 5

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 3/33
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=33)
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Blood pressure systolic increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Shire's agreements with investigators vary. All agreements provide Shire the right to embargo communications regarding trial results prior to public release for a period ≤180 days from the time submitted to Shire for review. Shire does not prohibit publication, but can require the removal of confidential information (excluding trial results) and can request postponement of a single-center publication until after disclosure of the trial's multi-center publication.